CLINICAL TRIAL: NCT06498869
Title: The Effect of Ketamine on Sleep Quality in Patients Undergoing Colonoscopy: A Prospective, Randomized, Controlled, Double-Blind Study
Brief Title: The Effect of Ketamine on Sleep Quality in Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KSH-ANREA-BG-02
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sleep
Keywords: Sleep Quality; Ketamine; Sleep; Sleep Habits; Anesthesia; Sedation; Colonoscopy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Our participants will be randomized into two separate groups. One group will receive midazolam and propofol, which will be our control group. The other group will receive ketamine in addition to midazolam and propofol during the procedure.
Who Masked: Participant, Investigator
Masking Description: Randomization will be conducted by an independent researcher (AY) using computer software and will be securely stored in sealed envelopes. An independent researcher (AŞ) will open the envelope 30 minutes prior to the procedure. The researcher administering anesthesia and the researcher conducting patient follow-ups and assessments (BG) will be blinded to each other. The participants will also be unaware of their assigned study group. Consequently, both the participants and the researcher assessing sleep quality (BG) will be blinded to the treatment administered. The study will be designed as a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Active Comparator): This group will receive ketamine (0.25-0.50 mg/kg) in addition to midazolam and propofol during the colonoscopy procedure
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj
- Control Group (No Intervention): For this group, midazolam and propofol will be administered during the colonoscopy procedure. Ketamine will not be administered additionally.

INTERVENTIONS:
Drug: Ketamine Hcl 50Mg/Ml Inj — This group will be administered ketamine (0.25-0.50 mg/kg)
  Other Names: Ketalar, Registry Number: 690G0D6V8H, Unique ID D007649
  Arms: Ketamine Group

SUMMARY:
Sedation typically begins with 2 mg of midazolam (0.025-0.1 mg/kg), followed by propofol given initially at 0.5-1.0 mg/kg bolus doses, with additional 0.25-0.5 mg/kg boluses as needed every 1-3 minutes to maintain sedation. Depending on clinical judgment, ketamine may be added to minimize propofol doses due to its minimal respiratory depression effects, administered at 0.25-0.50 mg/kg.

In the study protocol, participants undergo comprehensive assessments using the Pittsburgh Sleep Quality Index, Hospital Anxiety and Depression Scale, Numeric Rating Scale for Sleep Quality, and Richards Campbell Sleep Questionnaire on the procedure day, conducted in person.

Participants are randomized into two groups: one receiving midazolam and propofol (control group), and the other receiving ketamine in addition to midazolam and propofol.

Procedure duration and medication doses are meticulously recorded. Post-procedure, patients with a Modified Aldrete Score of 10 are transferred to the recovery unit. Participant data are documented, with follow-up conducted via phone 7 days post-procedure. Participants are reassessed using the aforementioned scales after the procedure, concluding the initial follow-up. The effects of ketamine on sleep quality will be evaluated by comparing the values of the mentioned scales before and after the procedure.

DETAILED DESCRIPTION:
During colonoscopy procedures, routine procedural sedation and analgesia are typically administered due to expected severe discomfort and pain. Sedation is administered by anesthesiologists using various medications according to established clinical guidelines, such as those outlined by the Turkish Society of Anesthesiology and Reanimation. Typically, an initial dose of 2 mg of midazolam (0.025-0.1 mg/kg) is administered, followed by propofol. Propofol is initially given at a bolus dose of 0.5-1.0 mg/kg, followed by additional bolus doses of 0.25-0.5 mg/kg at intervals of 1-3 minutes as required to achieve and maintain sedation. Depending on clinical judgment, some clinicians may supplement with ketamine, known for its minimal respiratory depression effects, to reduce propofol dosage. Ketamine is administered at doses of 0.25-0.50 mg/kg for this purpose. All medications are administered intravenously, aiming for a moderate sedation scale of 1-3 (TARD Non-operating Room Anesthesia Practice Guidelines, March 2022, page 17).

In the study protocol, participants will undergo the following procedures based on these guidelines.

Participants who consent to participate in the study will undergo assessment using the Pittsburgh Sleep Quality Index, Hospital Anxiety and Depression Scale, Numeric Rating Scale for Sleep Quality, and Richards Campbell Sleep Questionnaire on the day of the procedure. This assessment will be conducted in person.

Participants will be randomized into two groups. One group will receive midazolam and propofol, constituting the control group. The other group will receive ketamine in addition to midazolam and propofol during the procedure.

The duration of the procedure and total medication doses will be documented. After the procedure, patients achieving a Modified Aldrete Score of 10 will be discharged to the recovery unit (TARD Non-operating Room Anesthesia Practice Guidelines, March 2022, page 17).

Data on participants will be recorded, and they will be contacted by phone 7 days post-procedure.

Participants will undergo reassessment using the Pittsburgh Sleep Quality Index, Hospital Anxiety and Depression Scale, Numeric Rating Scale for Sleep Quality, and Richards Campbell Sleep Questionnaire scales after the procedure.

Following this assessment, participant follow-up will conclude. The effects of ketamine on sleep quality will be evaluated by comparing the values of the mentioned scales before and after the procedure.

Participants will be randomized into the Ketamine Group and Control Group in a 1:1 ratio. Randomization will be conducted using computer software by an independent researcher (AY). Randomization will be securely stored in sealed envelopes. An independent researcher (AŞ) will open the envelope 30 minutes prior to the procedure. The researcher administering anesthesia and the researcher conducting participant follow-ups and assessments (BG) will remain blinded to each other. Participants and the researcher assessing sleep quality (BG) will be unaware of the treatment administered to participants. The study is designed as a double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study
* Patients undergoing colonoscopy procedures
* Patients classified as ASA 1-2
* Male and female patients aged 18-65 years

Exclusion Criteria:

* Patients who decline to participate in the study
* Patients allergic to ketamine, propofol, and midazolam
* Patients with acute or chronic pain
* Patients diagnosed with psychiatric disorders
* Patients using antidepressants or sleep medications
* Patients with sleep disorders
* Patients with a history of oncological diseases
* Patients experiencing complications related to colonoscopy procedures
* Patients experiencing complications related to anesthesia administration
* Patients with a body mass index (BMI) >30 kg/m²
* Patients with cognitive impairment or communication issues
* Pregnant and postpartum patients
* Patients with sleep apnea syndrome
* Patients with uncontrolled hypertension (Blood Pressure >180/110 mmHg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Effects of Ketamine on Sleep Quality Scores | Postoperative at 7.day
  Ketamine, a dissociative anesthetic commonly used in medical and veterinary settings, has shown potential benefits for sleep quality, particularly in individuals with chronic pain or depression. Its primary mechanism involves blocking NMDA receptors in the brain, which not only provides anesthesa and pain relief but also impacts brain regions responsible for regulating sleep. Pittsburgh sleep quality index 0-21. RICHARD CAMPBELL sleep quality 0-100.SLEEP QUALITY NUMERICAL RATING SCALE 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: BEDİRHAN GÜNEL, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request can be made to obtain patient data from the institution. Data will not be shared by the researchers.

REFERENCES:
- [Background] Yang Y, Zhang Y, Zhou G, Yang Z, Yan H, Zhang J. Efficacy of epidural esketamine on postoperative sleep quality after laparoscopic and robotic lower abdominal surgeries: a study protocol for randomised, double-blind, controlled trial. BMJ Open. 2024 Feb 27;14(2):e081589. doi: 10.1136/bmjopen-2023-081589. PMID 38417951
- [Background] Cui M, Xing T, Zhao A, Zheng L, Zhang X, Xue H, Wu Z, Wang F, Zhao P. Effects of intraoperative sodium oxybate infusion on post-operative sleep quality in patients undergoing gynecological laparoscopic surgery: A randomized clinical trial. J Clin Anesth. 2024 May;93:111349. doi: 10.1016/j.jclinane.2023.111349. Epub 2023 Dec 1. PMID 38039631
- [Background] Qiu Y, Hou H, Zhang J, Wang X, Wang L, Wu Y, Deng L. The effect of preoperative sleep quality on the target plasma concentration of propofol and postoperative sleep in patients undergoing painless gastroscopy. BMC Anesthesiol. 2023 Jan 7;23(1):9. doi: 10.1186/s12871-022-01957-2. PMID 36609213